CLINICAL TRIAL: NCT02574715
Title: A Cross-sectional, Observational Study to Assess Quality of Life and Satisfaction of Young Women (Aged 18-29) Following 6 (±1) Months Using Jaydess® as Their Contraceptive Method - The JULIA Study.
Brief Title: An Observational Study to Assess Quality of Life and Satisfaction of Young Women (Aged 18-29) Following 6 (±1) Months Using Jaydess as Their Contraceptive Method
Acronym: JULIA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18096
Record Dates: First submitted 2015-09-21; First posted 2015-10-14 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Quality of Life
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Levonorgestrel (Jaydess, BAY86-5028): women aged 18 to 29 years following 6 (±1) months of Jaydess® use as their contraceptive method.
  Interventions: Drug: Levonorgestrel (Jaydess, BAY86-5028)

INTERVENTIONS:
Drug: Levonorgestrel (Jaydess, BAY86-5028) — Intrauterine delivery system Jaydess (13.5 mg levonorgestrel)

SUMMARY:
This is a cross-sectional, multicenter observational study to assess quality of life in young Spanish women (aged 18 to 29) who use Jaydess® as their contraceptive method. The study will be conducted in standard clinical practice conditions at the private gynecology clinics and during a single study visit.

Approximately 1,200 women who have been using the intrauterine delivery system (IUS) Jaydess® as their contraceptive method of choice for 6 (±1) months will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 29 years.
* Women who have been using Jaydess as their contraceptive method for 6 (±1) months.
* Women who have no comprehension, reading or writing challenges.
* Women who have given informed consent in writing.

Exclusion Criteria:

* Contraindication to the use of Jaydess.
* Prescription of Jaydess® for non-contraceptive medical reasons.
* Women who are considered to be unsuitable to take part in the study by the investigator (e.g., poor understanding of the study characteristics, uncooperative, etc.).
* Women who are currently taking part in any clinical trial.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 1,200 women aged 18 to 29 will be consecutively included in this study as they present at private gynecology clinics. Subjects must have been using the Jaydess intrauterine delivery system as their contraceptive of choice for a period of 6 (±1) months.
  The study population may be stratified into subsets to assess and identify differences in the subjects' quality of life, social and demographic characteristics, contraception characteristics, satisfaction, perceived benefits of Jaydess and bleeding pattern features.
Sampling Method: Non-Probability Sample
Enrollment: 1039 (Actual)
Dates: Start 2015-09-18 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-09-28 (Actual)

PRIMARY OUTCOMES:
Quality of life as determined using the SEC-QoL scale | At the single visit
  SEC-QoL (Spanish Contraception Society Quality of Life Questionnaire) is to assess the impact of contraceptive methods on health-related quality of life in women.

SECONDARY OUTCOMES:
Age (years) | At the single visit
Marital Status | At the single visit
Place of Birth | At the single visit
Place of residence (province, town, city or rural area) | At the single visit
Educational level (primary, secondary or higher education) | At the single visit
Employment (working outside the home, working from home, unemployed, student) | At the single visit
Maternity status (has children or plans to have children) | At the single visit
Frequency attending this physician's clinic for family planning purposes | At the single visit
History of type of contraceptive use | At the single visit
History of duration of contraceptive use | At the single visit
Prescription of Jaydess (date) | At the single visit
Benefits perceived on ease and comfort of use by means of a structured interview (Yes, No) | At the single visit
  This will be assessed by a structured interview during which the subject will be asked a number of questions by her gynecologist with answers (Yes or No): Indicate the advantages of Jaydess (select all that apply): comfort, avoid forgetfulness, reversibility, long duration, contraception cost, ease of use, safety, reduction in the duration and amount of bleeding, regulation of menstrual cycle, decreased menstrual pain, immediate contraceptive activity, high efficacy.
Global assessment of the insertion by means of a structured interview for pain questions (any, slight, moderate, severe) | At the single visit
Global assessment of the insertion by means of a structured interview for times questions | At the single visit
Global assessment of the insertion (acceptable without discomfort, with a few of minimal discomfort or with an enormous discomfort and unacceptable) | At the single visit
Global satisfaction with Jaydess, using a structured questionaire | At the single visit
  Satisfaction with Jaydess will be assessed using a structured questionnaire. The ease of use and impact on activities of daily living dimensions will be assessed on 3 items (ease and comfort of use, impact on activities of daily living and sexuality) for each dimension, each one with a 5-item Likert-like scale (where 1 = extremely unsatisfied and 5 = extremely satisfied).
Bleeding pattern features, using a questionnaire to compare current bleeding versus bleeding before the insertion of Jaydess as recalled | At the single visit

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Spain